CLINICAL TRIAL: NCT07156747
Title: Evaluate the Impact of Dynamic Video Education Versus Static Images and Verbal Instruction on Pain Perception and Anxiety in Patients Undergoing Transrectal Ultrasound-guided Prostate Biopsy (TRUS-Bx).
Brief Title: The Impact of Video Education on Pain and Anxiety in Patients Undergoing Transrectal Ultrasonography-Guided Prostate Biopsy
Acronym: TRUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Fatih SANDIKCI, Dr. Fatih SANDIKCI, Urology Specialist, Principal Investigator, Ankara Etlik City Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AESH-U-FS-01
Record Dates: First submitted 2025-08-02; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Prostate Biopsy; Anxiety
Keywords: Prostate Biopsy; Video Education; Pain Perception; Anxiety; Patient Preparation
MeSH Terms: conditions — Prostatic Neoplasms; Anxiety Disorders | interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: Participants were categorized into three groups. The control group received verbal information regarding the biopsy procedure. The film Group received a same verbal explanation and viewed a brief film regarding TRUS-Bx sourced from a widely utilized video-sharing platform. The picture group received verbal information accompanied by still photographs depicting the biopsy procedure. Participants in this trial were not randomized. Rather, they were allocated to groups according to their socioeconomic level. This was implemented to deliver education tailored to each patient's background and comprehension. All teaching initiatives were administered by the same qualified urology nurse to maintain consistency. A panel of urologists pre-selected the video and graphic elements for clarity, accuracy, and educational value.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Experimental): The control group received verbal information regarding the biopsy procedure.
  Interventions: Other: Visual Analog Scale; Other: State-Trait Anxiety Inventory
- Video Group (Experimental): The Video Group viewed a brief video about TRUS-Bx that was sourced from a frequently utilized video-sharing platform.
  Interventions: Other: Visual Analog Scale; Other: State-Trait Anxiety Inventory; Other: Video
- Image Group (Experimental): The image group (Image Group) was provided with information and still images that depicted the biopsy procedure.
  Interventions: Other: Visual Analog Scale; Other: State-Trait Anxiety Inventory; Other: Image

INTERVENTIONS:
Other: Visual Analog Scale — The Visual Analog Scale (VAS) is a linear instrument employed to measure perceived pain intensity, spanning from 0 (indicating no pain) to 10 (representing the most severe pain), where patients indicate the level that most accurately represents their experience.
Other: State-Trait Anxiety Inventory — The STAI is a self-administered questionnaire with two parts: STAI-1 measures state anxiety, representing a transient emotional state triggered by a particular circumstance, while STAI-2 examines trait anxiety, denoting a consistent predisposition to experience anxiety across diverse situations.
Other: Video — watching video on Digital Platfrom (for example, Youtube)
  Arms: Video Group
Other: Image — Prostate biopsy information with images
  Arms: Image Group

SUMMARY:
This study aimed to assess the impact of dynamic video education versus static images and verbal instruction on pain perception and anxiety in patients undergoing transrectal ultrasound-guided prostate biopsy (TRUS-Bx).

Participants were allocated to three groups: control (verbal information), video (verbal information accompanied by dynamic video), and image (verbal information supplemented by static images). Pain intensity was quantified utilizing the Visual Analog Scale (VAS), while anxiety was evaluated with the State-Trait Anxiety Inventory (STAI) prior to and following the surgery.

DETAILED DESCRIPTION:
Prostate cancer is among the most common malignancies diagnosed globally and constitutes the second highest cause of cancer-related mortality in males. Timely identification is crucial for enhancing clinical results, directing suitable therapy alternatives, and ultimately elevating survival rates. Transrectal ultrasound-guided prostate biopsy (TRUS-Bx) is the definitive diagnostic method for acquiring tissue samples from suspected prostate lesions. This method is preferred because of its comparatively low expense, extensive accessibility, and significant diagnostic efficacy.

Although categorized as a minimally invasive technique, TRUS-Bx can induce significant psychological anguish in patients. Pre-procedural anxiety is prevalent and can stem from various factors: dread of discomfort related with the biopsy, concern regarding a possible cancer diagnosis, and lack of familiarity or misunderstanding about the biopsy procedure. This worry is not solely an emotional concern; it can negatively impact physiological metrics such as blood pressure and heart rate, heighten the perceived discomfort during the surgery, and diminish patient compliance. Furthermore, elevated anxiety levels are associated with diminished patient satisfaction and can adversely affect patients' readiness to pursue essential medical procedures in the future, potentially resulting in long-term health repercussions.

Reducing preoperative anxiety is essential for patient-centered treatment in procedural medicine. Effective educational interventions have demonstrated the capacity to alleviate anxiety by improving patient comprehension and establishing reasonable expectations. Conventional approaches encompass oral elucidations by healthcare professionals and printed pamphlets, whose efficacy fluctuates owing to disparities in literacy, attention, and retention among patients. Visual aids, particularly educational movies, provide a multimodal learning experience by integrating aural narrative with dynamic visuals, which may enhance understanding and engagement.

Prior studies on diverse medical procedures, including colonoscopy, endoscopy, and small surgical interventions, have shown that video-based teaching can markedly boost patients' understanding, alleviate anxiety, and improve overall satisfaction with the care experience. Nonetheless, despite the prevalent application of TRUS-Bx, there is a scarcity of data investigating the particular influence of video education in this domain. Moreover, it is uncertain whether dynamic video content (e.g., animated or actual procedural footage) provides benefits over static visuals or verbal information alone in mitigating anxiety and perceived pain associated with prostate biopsy.

Moreover, due to the growing accessibility of internet video platforms such as YouTube, individuals frequently pursue information autonomously before undergoing medical operations. Although this can empower patients, the quality and accuracy of such content fluctuate significantly, potentially affecting their psychological condition in unforeseen manners.

Research Aim

This study seeks to systematically assess the impact of pre-procedural video education regarding TRUS-Bx on patients' anxiety and subjective pain levels. The researchers aim to compare the impact of dynamic, detailed videos-akin to those found on popular platforms such as YouTube-with static image displays or traditional spoken therapy. The fundamental premise posits that exposure to extensive, dynamic video information before biopsy will adequately prepare patients by clarifying the technique, therefore alleviating psychological discomfort and enhancing their overall experience.

This study aims to clarify the function of video-based instructional aids in the clinical environment, intending to guide best practices for patient education and aid in the formulation of standardized procedures to enhance patient-centered outcomes in prostate cancer diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Men between 50 and 80 years of age
* Elevated prostate-specific antigen (PSA) levels and/or suspicious digital rectal examination (DRE) findings
* Literacy and comprehension

Exclusion Criteria:

* A history of previous prostate biopsy
* Cognitive or psychiatric disorders
* Using anxiolytic medications
* After being informed, declining to participate in the study

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Our study will be conducted on patients scheduled for prostate biopsy. Therefore, all participants are male.
Enrollment: 223 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
The importance of biopsy procedure information | Through study completion, an average of 1 year
  The research indicates that an increase in patients' anxiety-stress ratings will require the implementation of supplementary measures to notify patients prior to the treatment. Patients who decline the surgery may encounter delays in diagnosis and treatment, or these may be entirely omitted, owing to the visual information and videos acquired prior to the procedure. This study will additionally function as a reference for image alteration on digital platforms. By assessing the levels of anxiety and discomfort induced by visual and verbal input, modifications can be implemented in the information processes related to the procedure.
Assessment of pain intensity associated with the biopsy operation | Through study completion, an average of 1 year]
  The Visual Analog Scale (VAS) is a linear measurement tool used to assess perceived pain intensity, ranging from 0 (indicating no pain) to 10 (representing the most severe pain), where patients indicate the level that most accurately represents their experience. All measurements were conducted in a tranquil environment immediately prior to and following the biopsy process.
Evaluation of anxiety levels related to the biopsy procedure | Through study completion, an average of 1 year
  The STAI is a self-administered questionnaire with two elements: STAI-1 measures state anxiety, representing a transient emotional state elicited by a particular circumstance, while STAI-2 examines trait anxiety, signifying a consistent predisposition to experience anxiety across diverse situations. State-Trait Anxiety Inventory, Form 1 and Form 2 (STAI-1 and STAI-2). It is a Likert scale. The cumulative score derived from both measures runs from 20 (indicating mild anxiety) to 80 (indicating excessive anxiety). Diverse scoring methodologies are available for STAI-1 and STAI-2 scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tarhan H, Cakmak O, Unal E, Akarken I, Un S, Ekin RG, Konyalioglu E, Isoglu CS, Zorlu F. The effect of video-based education on patient anxiety in men undergoing transrectal prostate biopsy. Can Urol Assoc J. 2014 Nov;8(11-12):E894-900. doi: 10.5489/cuaj.2208. PMID 25553162
- [Result] Sheng LP, Han CQ, Nie C, Xu T, Zhang K, Li XJ, Xie XR, Lin R, Ding Z. Watching Videos of Colonoscopies and Receiving Interpretations Reduce Pain and Anxiety While Increasing the Satisfaction of Patients. Dig Dis Sci. 2021 Feb;66(2):541-546. doi: 10.1007/s10620-020-06186-6. Epub 2020 Mar 19. PMID 32193861
- [Result] Bujnowska-Fedak MM, Wegierek P. The Impact of Online Health Information on Patient Health Behaviours and Making Decisions Concerning Health. Int J Environ Res Public Health. 2020 Jan 31;17(3):880. doi: 10.3390/ijerph17030880. PMID 32023828
- [Result] Monteiro Grilo A, Ferreira AC, Pedro Ramos M, Carolino E, Filipa Pires A, Vieira L. Effectiveness of educational videos on patient's preparation for diagnostic procedures: Systematic review and Meta-Analysis. Prev Med Rep. 2022 Jul 5;28:101895. doi: 10.1016/j.pmedr.2022.101895. eCollection 2022 Aug. PMID 35855928
- [Result] Sefik E, Gunlusoy B, Eker A, Celik S, Ceylan Y, Koskderelioglu A, Basmaci I, Degirmenci T. Anxiety and depression associated with a positive prostate biopsy result: A comparative, prospective cohort study. Int Braz J Urol. 2020 Nov-Dec;46(6):993-1005. doi: 10.1590/S1677-5538.IBJU.2019.0719. PMID 32822128

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT07156747/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT07156747/ICF_001.pdf